## Smart digital denture conversion (SDDC), a technique for full arch immediate loading.

Document Date: October 27, 2023

The obtained data will be recorded, tabulated, and statistically analyzed using the Mann-Whitney U Test was used for comparison between the two groups. Statistics was done with IBM SPSS statistics v20. Data was presented as median and interquartile range.